CLINICAL TRIAL: NCT06588478
Title: A Phase 2, Open-Label, Randomized Study Evaluating the Efficacy and Safety of 3 Doses of Pirtobrutinib in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Who Previously Received Treatment With a Covalent Bruton Tyrosine Kinase Inhibitor
Brief Title: A Study Evaluating the Efficacy and Safety of Pirtobrutinib in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18877; 2024-515689-15-01 (EU CTIS Number); J2N-MC-JZNX (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib

STUDY DESIGN:
Masking Description: Part 2 is non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pirtobrutinib Standard Dose (Dose 1)-Part 1 (Active Comparator): Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Dose 2-Part 1 (Experimental): Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Dose 3-Part 1 (Experimental): Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Standard Dose-Part 2 (Experimental): Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered Orally.

SUMMARY:
The main purpose of Part 1 of this study is to assess the efficacy and safety of 3 dose levels of Pirtobrutinib in participants with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), who have received 1-3 lines of treatment including a covalent Bruton tyrosine kinase (BTK) inhibitor. The purpose of Part 2 of this study is to evaluate pirtobrutinib monotherapy in participants with treatment-naïve CLL/SLL with 17p deletions. Participation in Part 1 is expected to last approximately 3 years. Participation in Part 2 is expected to last up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of CLL/SLL as defined by iwCLL 2018 criteria.
* Part 1: Have received prior CLL/SLL treatment
* Have received at least 1, but not more than 3 lines of prior treatment for CLL/SLL
* Have received a covalent BTK inhibitor
* Part 2: Have received no prior treatment for CLL/SLL

  * Part 1 - Known 17p deletion status (positive or negative)
  * Part 2 - Must have 17p deletion (positive)
* Have a requirement for therapy consistent with iwCLL 2018 criteria for initiation of therapy
* Capable of swallowing oral study medication.
* Have an Eastern Cooperative Oncology Group Performance Status (ECOG) score of 0 to 2.

Exclusion Criteria:

* Have received prior treatment with a BTK degrader or a noncovalent BTK inhibitor
* Have a history of greater than or equal to (>=) Grade 3 bleeding due to treatment with a BTK inhibitor
* Have known or suspected Richter's transformation
* Have known or suspected history of central nervous system involvement by CLL/SLL
* Previous or concurrent cancer distinct from CLL/SLL within 3 years before randomization. Exceptions may occur with documented sponsor approval. Examples include:

  * nonmelanoma skin cancer or lentigo malignant melanoma
  * cervical carcinoma in situ
  * localized prostate cancer undergoing active surveillance, and
  * localized (for example, lymph node negative) breast cancer with no evidence of active disease present for more than 3 years. Individual may be receiving adjuvant hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Baseline up to 3 years
  Overall response rate is defined as the proportion of participants who achieve the best overall response at or before the initiation of subsequent anticancer therapy of CR, CRi, nPR, or PR. ORR will be assessed using International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 response criteria.

SECONDARY OUTCOMES:
Duration of Response | Baseline up to 3 years
  Duration of response is defined as the time from the date of the first documented CR, CRi, nPR, or PR to disease progression (per iwCLL 2018) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (134):
- United States (22):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - City of Hope National Medical Center, Duarte, California
  - City of Hope National Medical Center, Irvine, California
  - Palo Alto Medical Foundation Research Institute (PAMFRI), Palo Alto, California
  - Stanford Cancer Center, Palo Alto, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - City of Hope National Medical Center, Atlanta Cancer Center, Newnan, Georgia
  - Mission Cancer + Blood, Waukee, Iowa
  - Saint Elizabeth Medical Center Edgewood, Edgewood, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Clinical Research Alliance, Westbury, New York
  - East Carolina University, Greenville, North Carolina
  - Williamette Valley Cancer Institute & Research Center, Eugene, Oregon
  - Cancer Care Associates Of York, York, Pennsylvania
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - USO-Texas Oncology-Central/South Texas, Austin, Texas
  - Sarah Cannon Research Institute/SCRI, The Woodlands, Texas
  - USO-Virginia Oncology Associates, Hampton, Virginia
- Australia (10):
  - Flinders Medical Centre, Adelaide
  - Bankstown-Lidcombe Hospital, Bankstown
  - Box Hill Hospital, Box Hill
  - Coffs Harbour Health Campus, Coffs Harbour
  - Royal Hobart Hospital, Hobart
  - ICON Cancer Centre - Kurralta Park, Kurralta Park
  - Latrobe Regional Health, Traralgon
  - Calvary Mater Newcastle, Waratah
  - The Perth Blood Institute - West Perth, West Perth
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (9):
  - Institut Jules Bordet, Anderlecht
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - UZ Gent, Ghent
  - Groupe Jolimont, La Louvière
  - UZ Leuven, Leuven
  - Clinique Saint Pierre, Ottignies
  - AZ Delta vzw, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - CHR Verviers - La Tourelle, Verviers
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie
  - Saskatoon Cancer Centre, Saskatoon
- Czechia (4):
  - Fakultní nemocnice Brno Bohunice, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Odense Universitetshospital, Odense
- France (6):
  - Centre Hospitalier d'Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre, Caen
  - Centre Hospitalier du Mans, Le Mans
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace - Hôpital Emile Muller, Mulhouse
  - Centre Antoine-Lacassagne, Nice
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
- Germany (6):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - MV-Zentrum für Onkologie und Hämatologie, Cologne
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - OSP Göttingen, Göttingen
  - Onkologisches Ambulanzzentrum Hannover, Hanover
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz
- Greece (4):
  - Evangelismos General Hospital of Athens, Athens
  - Attikon General University Hospital, Chaïdári
  - G. Papanikolaou General Hospital, Thessaloniki
  - General Hospital of Athens "Laiko", Αthens
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Dél-Pesti Centrumkórház, Budapest
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Italy (10):
  - A.O.U.C. Policlinico di Bari, Bari
  - Azienda Ospedaliero Universitaria S.Anna, Cona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Azienda Ospedale - Università Padova, Padua
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO, Palermo
  - AO Santa Maria della Misericordia, Perugia
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- Poland (5):
  - IN VIVO, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - AIDPORT Sp. z o.o., Skórzewo
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- Romania (6):
  - Fundeni Clinical Institute, Bucharest
  - Spitalul Clinic Colțea, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - Institutul Regional de Oncologie, Iași
  - Ovidius Clinical Hospital OCH, Ovidiu
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
  - Univerzitna Nemocnica L. Pasteura Kosice, Košice
  - Univerzitna nemocnica Martin, Martin
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
- Spain (16):
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet Del Llobregat
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Costa del Sol, Marbella
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Turkey (Türkiye) (9):
  - Sakarya University School of Medicine, Adapazarı
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Memorial Antalya Hospital, Antalya
  - Yeditepe Üniversitesi Koşuyolu Hastanesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Kocaeli Üniversitesi, İzmit
  - VM Medical Park Mersin Hastanesi, Mersin
  - Ondokuz Mayıs Universitesi, Samsun
- United Kingdom (9):
  - Heartlands Hospital, Birmingham
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Northwick Park Hospital, Harrow
  - St James's University Hospital, Leeds
  - Lincoln County Hospital, Lincoln
  - Clatterbridge Cancer Centre - Liverpool, Liverpool
  - Hammersmith Hospital, London
  - Maidstone Hospital, Maidstone
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/